CLINICAL TRIAL: NCT05225831
Title: Safety and Efficacy of CD19/CD22 Dual Targeted CAR-T Cell Therapy in Patients With R/R B-Cell Acute Lymphoblastic Leukemia
Brief Title: Safety and Efficacy of CD19/CD22 Dual Targeted CAR-T Cell Therapy in R/R B-Cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL19+22 for B-ALL
Record Dates: First submitted 2022-01-11; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: CD19+ and CD 22+ B-ALL
Keywords: CD19; CD22; B-ALL; CAR-T
MeSH Terms: interventions — CF regimen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SL19+22 CAR-T (Experimental): Eligible patients will be treated with SL19+22 CAR-T.
  Interventions: Biological: Autologous CD19/CD22 Chimeric Antigen Receptor T-cells; Drug: Cyclophosphamide,Fludarabine

INTERVENTIONS:
Biological: Autologous CD19/CD22 Chimeric Antigen Receptor T-cells — A single infusion of CD19 and CD22 CAR-T cells.
  Other Names: SL19+22 CAR-T
Drug: Cyclophosphamide,Fludarabine — Given

SUMMARY:
This is an open, single-arm, prospective clinical study to evaluate the safety and efficacy of anti CD19 and CD22 CAR-T cell in the treatment of R/R B-ALL.

DETAILED DESCRIPTION:
CD19-directed CAR-T cell therapy has shown promising results in the treatment of relapsed/refractory B-cell acute lymphoblastic leukemia. CD19 and CD22 are proteins usually expressed on the surface of the B leukemia cells. The dual-CARs enables the T-cells to recognize and kill the tumor cell through recognition of CD19 and CD22.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent and be willing and able to comply with the visit, treatment regimen, laboratory examination and other requirements of the study as stipulated in the trial flow chart;
2. A definite diagnosis of B-cell Lymphocyte Leukemia, which meets any of the following criteria: Relapsed : a) relapsed within 12 months after first remission;Refractory: a) no remission after six weeks of induction therapy or no remission after two courses of induction therapy; b) relapsedafter CR for 2 or more times; c) The first relapse after chemotherapy and no remission after at least one salvage treatment; c) relapsed after hematopoietic stem cell transplantation;
3. ECOG Scores: 0~2
4. CD19 positive and CD22 positive were detected by immunohistochemistry or flow cytometry;
5. Estimated survival time>3 months;
6. Peripheral blood mononuclear immune cells must be collected at least 2 weeks after the last radiotherapy or systemic treatment.
7. For patients with only extramedullary recurrence of B-ALL, there must be at least one assessable lesion.

Exclusion Criteria:

1. Serious cardiac insufficiency；
2. Has a history of severe pulmonary function damaging;
3. Presence of other malignant tumors.
4. Presence of active fungal, bacterial, viral, or other infection requiring IV antibiotics for management.
5. Presence of other severe autoimmune diseases or immunodeficiency disease;
6. Patients with active hepatitis B or hepatitis C([HBVDNA+]or [HCVRNA+]);
7. Known positive serology for human immunodeficiency virus (HIV) or syphilis。
8. Has a history of serious allergies on biological products (including antibiotics);
9. Female patients who are under pregnancy and/or lactation, or planing on pregnancy for the next 12 months.
10. Any other situations that the researchers believe will affect the results of the study.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | up to 28 days
  To evaluate the possible adverse events that could occurred within the first month post SL19+22 infusion, including symptoms such as cytokine release syndrome and neurotoxicity.
Efficacy: Remission Rate | Up to 3 months
  Remission Rate includes complete remission(CR)、CR with incomplete blood count recovery(CRi)、No remission(NR)

SECONDARY OUTCOMES:
Efficacy:duration of response (DOR) | 24 months post CAR-T cells infusion
  Duration of response
Efficacy: progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of CD19 and CD22 CAR- T cells in the genomes of peripheral blood mononuclear cell (PBMC) by quantitative Real-time PCR (qPCR).
Cytokine release | First month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD&MD, Principal Investigator — Beijing Lu Daopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Langfang, Hebei, China